CLINICAL TRIAL: NCT05674656
Title: Phase 1/2 Study of Switching to Fixed Dose Combination Dolutegravir/Rilpivirine Among Virologically Suppressed Children, 6 to Less Than 12 Years of Age, Living With HIV-1
Brief Title: Pharmacokinetics, Safety, Tolerability of Dolutegravir/Rilpivirine in Pediatrics
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205868; 2022-000829-24 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2023-01-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections
Keywords: Dolutegravir; Rilpivirine; JULUCA
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; dolutegravir, rilpivirine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dolutegravir(DTG)/Rilpivirine (RPV) (Experimental)
  Interventions: Drug: Dolutegravir/Rilpivirine FDC

INTERVENTIONS:
Drug: Dolutegravir/Rilpivirine FDC — Dolutegravir/Rilpivirine will be administered.
  Other Names: JULUCA

SUMMARY:
The purpose of this study is to provide data on the pharmacokinetic (PK), safety, tolerability, efficacy and acceptability of this fixed dose combination (FDC) single tablet 2-drug regimen for virologically suppressed (HIV-1 RNA [Ribonucleic Acid] < 50 [cells per milliliter] c/mL) children 6 to less than 12 years of age, weighing at least 25 kilogram (kg).

ELIGIBILITY:
Inclusion Criteria:

* Human immuno virus Type-1 (HIV-1) infected child 6 years to less than 12 years of age at the time of signing the informed consent form .
* Body weight greater than or equal to 25 kilogram (kg) at entry.
* Confirmed HIV-1-infection
* Participant has taken the same Antiretroviral therapy (ART) regimen in the 6 months (180 days) prior to Screening, as determined by the site investigator based on participant/parent/guardian report and available medical records.
* Has a plasma HIV-1 Ribonucleic Acid (RNA) result less than 50 copies/mL at Screening
* Has at least one documented plasma HIV-1 RNA result less than the lower limit of detection of the assay from a specimen collected in the 6-12 months (180-365 days) prior to Screening OR Has at least one documented plasma HIV-1 RNA result less than the lower limit of detection of the assay from a specimen collected less than 6 months (within 179 days) prior to entry and at least one documented plasma HIV-1 RNA result less than the lower limit of detection of the assay from a specimen collected in the 12-18 months (365-545 days) prior to Screening
* For participants of reproductive potential (defined as having reached menarche), not pregnant based on testing performed at Screening (i.e., from a specimen collected within 30 days prior to entry) and at Baseline/Day 1.
* For participants of reproductive potential who are engaging in sexual activity that could lead to pregnancy, willing to use two methods of contraception while receiving study drug and for approximately one month after permanently discontinuing study drug, based on participant/parent/guardian report at entry.
* For participants of reproductive potential, not breastfeeding based on participant/parent/ guardian report at Baseline/Day 1.

Exclusion Criteria:

* Documented resistance (ever) to Non-nucleoside reverse transcriptase inhibitors (NNRTIs) or integrase inhibitors
* Documented HIV-1 RNA result greater than or equal to the lower limit of detection of the assay based on a specimen collected in the 12 months (365 days) prior to Screening
* Any change (ever) of any Antiretroviral (ARV) agent due to virologic failure, as determined by the site investigator based on participant/parent/guardian report and available medical records
* Has a history (ever) of allergy to DTG, RPV, or any other component of JULUCA as determined by the site investigator based on participant/parent/guardian report and available medical records.
* Has a history (ever) of congestive heart failure, symptomatic arrhythmia, or any clinically significant cardiac disease as determined by the site investigator based on participant/ parent/guardian report and available medical records
* Has a history (ever) of unstable liver disease (defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) as determined by the site investigator based on participant/parent/guardian report and available medical records
* Has any of the following as determined by the site investigator based on participant/ parent/guardian report and available medical records: Current clinical evidence of pancreatitis; Currently active AIDS-defining (WHO Clinical Stage 4) opportunistic infection; Currently active TB and/or current rifamycin-containing TB treatment.
* Has an anticipated need for any HCV therapy during the first 24 weeks of study and for HCV therapy based on interferon or any drugs that have a potential for adverse drug: drug interactions with study treatment throughout the entire study period.
* Receipt of the following as determined by the site investigator based on participant/ parent/guardian report and available medical records: Any investigational agent within 90 days prior to entry; Any prohibited medication within 30 days prior to entry; Any medication with a known risk of Torsades de Pointes within seven days prior to entry
* Receipt (ever) of an ART regimen that included both DTG and RPV, as determined by the site investigator based on participant/parent/guardian report and available medical records
* Any ≥ grade 3 result for the following based on grading per the Division of Acquired Immunodeficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events: Haemoglobin (<8.5 gram per deciliter [g/dL] or <5.25 millimoles per liter [mmol/L]); Absolute neutrophil count (<600 cells/mm^3 or <0.600 x 109 cells/L); Platelet count (<50,000cells/mm^3 or <50.00 x 109 cells/L); Estimated glomerular filtration rate (eGFR: <60ml/min/1.73m^2); ALT (≥5.0 x Upper limit of Normal [ULN]); Aspartate Aminotransferase (AST) (≥5.0 x ULN)
* Has the following combination of laboratory test results at screening: Alanine transaminase [ALT] greater than or equal to 3 x ULN and total bilirubin greater than or equal to 1.5 x ULN and direct bilirubin greater than 35% of total bilirubin
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening.
* QTc >450 milliseconds (msec) at Screening
* Severe acute malnutrition (Body Mass Index [BMI] for age <-3 or nutritional oedema)
* Has any documented or suspected clinically significant medical or psychiatric condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.
* The child is a ward of State or government.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-05-03 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC0-24h) of DTG | Up to Week 24
Area under the curve (AUC0-24h) of RPV | Up to Week 24
Number of Participants with Adverse Events (AEs) at Week 24 | At Week 24
Number of Participants with Grade 3 or higher AEs at Week 24 | At Week 24
Number of Participants with Grade 3 or higher AEs assessed as related to study drug at Week 24 | At Week 24
Number of Participants with Fatal AEs assessed as related to study drug at Week 24 | At Week 24
Number of Participants with Serious Adverse Events (SAEs) assessed as related to study drug at Week 24 | At Week 24
Number of Participants with AEs assessed as related to study drug that led to permanent discontinuation of study drug at Week 24 | At Week 24

SECONDARY OUTCOMES:
Proportion of Participants with HIV-1 RNA less than 50 copies per milliliter (c/mL) | At Week 24 and 48
Cluster of differentiation 4 (CD4+) Cell Count | At Week 24 and 48
Percentage of CD4+ Cell Count | At Week 24 and 48
Number of Participants with Adverse Events (AEs) at Week 48 | At Week 48
Number of Participants with Grade 3 or higher AEs at Week 48 | At Week 48
Number of Participants with Grade 3 or higher AEs assessed as related to study drug at Week 48 | At Week 48
Number of Participants with Fatal AEs assessed as related to study drug at Week 48 | At Week 48
Number of Participants with Serious Adverse Events (SAEs) assessed as related to study drug at Week 48 | At Week 48
Number of Participants with AEs assessed as related to study drug that led to permanent discontinuation of study drug at Week 48 | At Week 48
Minimum drug concentration (Cmin) of DTG | Up to Week 24
Cmin of RPV | Up to Week 24
Cmin of DTG at Week 4 Visit | Pre-dose, 1, 2, 4, 5, 6, 10 and 24 hours (h) post-dose at Week 4
Cmin of RPV at Week 4 Visit | Pre-dose, 1, 2, 4, 5, 6, 10 and 24 hours (h) post-dose at Week 4
Concentration of HIV-1 RNA | Baseline (Day 1), Week 4, 8, 12, 16, 20, 24, 36 and 48
Number of Participants with HIV-1 Genotype at the time of Virologic failure (HIV-1 RNA greater than or equal to 200 copies/mL) | Baseline (Day 1) and up to Week 48
Number of Participants with HIV-1 Phenotype at the time of Virologic failure (HIV-1 RNA greater than or equal to 200 copies/mL) | Up to Week 48
Number of Participants with HIV-1 genotypes at Baseline, Week 24 and 48 | Baseline (Day 1), Week 24 and 48
Number of Participants with Acceptability to JULUCA | At Week 4, 24 and 48
Number of Participants with Adherence to JULUCA | At Week 4, 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (7):
- United States (7):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf